CLINICAL TRIAL: NCT03757494
Title: Cranial Electrotherapy Stimulation in the Treatment of Posttraumatic Stress Disorder: A Feasibility, Safety and Efficacy Study
Brief Title: Cranial Electrotherapy Stimulation in the Treatment of Posttraumatic Stress Disorder
Acronym: CES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Rustad, Principal Investigator, White River Junction Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1286051
Record Dates: First submitted 2018-10-17; First posted 2018-11-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: PTSD, Post Traumatic Stress Disorder
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Intervention Model Description: Using Alpha Stim
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Use of Alpha Stim (Experimental): Use of Alpha Stim Device
  Interventions: Device: Alpha Stim

INTERVENTIONS:
Device: Alpha Stim — Use of Alpha Stim Device

SUMMARY:
This is a research study that will look at how well a treatment called Cranial Electrotherapy Stimulation (CES) works for patients who struggle with symptoms of Posttraumatic Stress Disorder. Cranial Electrotherapy Stimulation is delivered using a device called Alpha-Stim®. This is a safe, non-invasive treatment that applies a low-level pulsed electric current through the brain using clip-on electrodes attached to the earlobes. Cranial Electrotherapy Stimulation treats conditions such as physical pain, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

1. To ensure participants can safely receive Alpha-Stim®, eligible participants must meet all established screening criteria for safety during Alpha-Stim® using a safety screener (as assessed during phone screen and medical records review). We are screening to access for metal. These are conservative measures require a patient not having the following (unless MRI-safe): Cardiac pacemaker, implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord. The patient would additionally be required to not have an implanted cardiac defibrillator;
2. Outpatients 18-70 years of age (inclusive);
3. Meet DSM-V criteria for PTSD (acute or chronic) at the time of the screening and/or baseline visit; symptoms.
4. Have a baseline score of "Moderately Ill" or worse on the CGI-S;
5. Be on a stable psychotropic regimen for at least 6 weeks prior to baseline, or no psychotropic medication at all (for at least 6 weeks prior to baseline), and be willing to maintain the current regimen and dosing for the duration of the study (unless medically necessary to make changes with notification of research staff);

(7) If female and of child bearing potential, agree to use an acceptable method of birth control for the duration of the study treatment period; (8) Be willing and able to comply with all study related procedures and visits; (9) Be capable of independently reading and understanding patient information materials and giving written informed consent.

-

Exclusion Criteria:

Participants will be excluded from participation if they meet any of the following:

1. Are pregnant or lactating or planning to become pregnant within the next three months;
2. Have a lifetime history of loss of consciousness due to head injury for greater than 10 minutes, or any lifetime history of loss of consciousness due to a head injury with documented evidence of brain injury (including brain atrophy);
3. Current (or past if appropriate) significant neurological disorder, or lifetime history of a) seizure disorder b) primary or secondary CNS tumors c) stroke or d) cerebral aneurysm;
4. Unstable medical illness, or, in the opinion of the investigator, significant absence of appropriate medical care;
5. Current Axis 1 primary psychotic disorder, or bipolar I disorder, active moderate/severe substance use disorders (within the last month as assessed by review of the medical records and veteran self-report, excluding nicotine/caffeine). Veterans on stable (>3 months), monitored opiate agonist therapy may be included at the investigator's discretion;
6. Past failed treatment with rTMS or ECT; any past treatment with deep brain stimulation or vagus nerve stimulation;
7. Have active suicidal intent or plan as detected on screening assessments, or in the Investigator's opinion, is likely to attempt suicide within the next six months;
8. Mental retardation or cognitive impairment
9. History of stroke, Parkinson's Disease, Multiple Sclerosis, or seizures
10. Current use of Transcutaneous electrical nerve stimulation (TENS) unit
11. Previous history of Alpha-Stim® use
12. Inability to read and write in English
13. Incapacity to make informed medical decisions for any reason
14. Pregnancy: Pregnant women are not eligible for the study. Women with potential for pregnancy will receive a pregnancy test provided by the VA prior to the study. Women of childbearing capacity are eligible for the study. Contraceptive plans will be discussed and if they are determined to be inadequate, the participant will be excluded from the study.
15. Presence of an implanted defibrillator or pacemaker device.
16. Demonstrate the presence of any other condition or circumstance that, in the opinion of the investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of Alpha-Stim® Cranial Electrotherapy Stimulation (CES) as a treatment for Posttraumatic Stress Disorder (PTSD). | 1 year
  We will deem the treatment feasible if ≥ 6 participants complete the protocol, based on completion of ≥ 60% treatments (3 out of 5 treatment days, weekly at home), and attending and completing ≥ 75% of the weekly assessments, including the week 1 baseline and week 4 treatment completion visit

SECONDARY OUTCOMES:
Safety of the Alpha-Stim® Cranial Electrotherapy Stimulation (CES) as a treatment for Posttraumatic Stress Disorder. | 1 year
  Safety and tolerability, we expect this treatment to be safe, based on the very few adverse events and no serious adverse events in the literature and relative safety when compared to current pharmacologic treatments (e.g., SSRIs and SNRIs) for PTSD.

OTHER OUTCOMES:
Efficacy of Alpha-Stim® Cranial Electrotherapy Stimulation (CES) as a treatment for Posttraumatic Stress Disorder. | 1 year
  Efficacy, while the study isn't powered for an efficacy trial, the initial screening to baseline pretreatment to post-treatment change in the magnitude of change in PTSD symptoms (as measured by the PCL-5) during Alpha-Stim® treatment using paired t-tests can be used to determine sample size and power calculations for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: James K Rustad, MD, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VAMC, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No